CLINICAL TRIAL: NCT06489821
Title: STereotactic Body Radiotherapy (SBRT) After oligoprogRession Metastatic Breast Cancer (STAR-B)
Brief Title: STereotactic Body Radiotherapy (SBRT) for Oligoprogressive Breast Cancer
Acronym: STAR-B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juravinski Cancer Center (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Principal Investigator, Elysia Donovan, Radiation Oncologist, Juravinski Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-B
Record Dates: First submitted 2023-11-16; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer; Oligoprogression
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic body radiotherapy (SBRT) plus continuation of first line systemic therapy (Experimental): SBRT in 5 or 2 (or 4) fractions for body and spine respectively over 2 weeks, while continuing first line systemic therapy
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Stereotactic body radiotherapy in 5 fractions (body) or 2 or 4 fractions (spine) plus continuation of first line systemic therapy

SUMMARY:
Recent advances in systemic therapy have facilitated improved progression-free survival (PFS) and treatment tolerability in metastatic breast cancer patients (MBC). Oligoprogression (OP) refers to progression limited to five or fewer sites in otherwise controlled systemic disease on a drug therapy. Stereotactic body radiotherapy (SBRT) has the potential to locally ablate resistant OP lesions that develop on a systemic treatment, and may consequently delay the need for change in drug therapy, delay time to chemotherapy and prolong PFS. This is a phase II trial of SBRT plus continuation of current systemic therapy line for OP MBC patients, to determine rate of delay of change in systemic therapy of at six months. PFS, time to chemotherapy and quality of life will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of progressive metastatic breast cancer on first line systemic therapy, including either hormone receptor positive, Her-2 negative (HR+/Her2-) on endocrine therapy + CDK4/6 inhibitor or Her-2 positive (hormone receptor positive or negative /Her2+) on Her2-targeted therapy regimens.
2. Progressive disease limited to "oligoprogression", defined as progression of 5 or fewer extra-cranial lesions with otherwise controlled systemic disease on current line of systemic therapy.
3. Patients must have previously controlled disease for at least six months on current systemic therapy
4. Deemed a candidate for stereotactic body radiotherapy (SBRT) to all OP lesions

Exclusion Criteria:

1. Requires change in systemic therapy line at the time of OP as determined by medical oncologist;
2. Progression on 2nd line or subsequent lines of therapy
3. Lacks CT or bone scan Imaging within previous 45 days;
4. Progression in >3 sites in the liver or lung;
5. Hormone positive disease on endocrine therapy only at time of enrollment;
6. Previous radiotherapy to same site or vicinity preventing definitive SBRT (e.g. within 5 cm);
7. Lesions deemed not amenable to SBRT due to large size or location;
8. Unacceptable fracture risk according to clinician judgement for bone lesions;
9. Brain metastasis or Spinal cord compression;
10. History of major radiosensitivity syndrome or contraindications to radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with change in systemic therapy | Six months
  Change in systemic therapy will occur with progression with the following criteria:
  1. Progression not amenable to further SBRT, including multifocal (>3) sites;
  2. Progression in lesion not amenable to further SBRT;
  3. Rapid progression such that treating medical oncologist believes change in therapy is warranted;
  4. Progression in location including, including visceral metastasis, such that treating medical oncologist believes change in therapy is warranted

SECONDARY OUTCOMES:
Progression-free survival | 3, 6, 12, 18, and 24 months
  Progression outside radiotherapy field per RECIST 1.1
Local progression | 3, 6, 12, 18, and 24 months
  Progression within a treated lesion per RECIST 1.1
Time to chemotherapy | 3, 6, 12, 18, and 24 months
  Initiation of cytotoxic therapy
Overall Survival | 3, 6, 12, 18, and 24 months
  Proportion of patients alive
CTCAE Toxicity | 3, 6, 12, 18, and 24 months
  common terminology criteria for adverse events 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Kyle McGowan, Study Director — Juravinski CC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Blackwell KL, Andre F, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Petrakova K, Hart LL, Villanueva C, Chan A, Jakobsen E, Nusch A, Burdaeva O, Grischke EM, Alba E, Wist E, Marschner N, Favret AM, Yardley D, Bachelot T, Tseng LM, Blau S, Xuan F, Souami F, Miller M, Germa C, Hirawat S, O'Shaughnessy J. Ribociclib as First-Line Therapy for HR-Positive, Advanced Breast Cancer. N Engl J Med. 2016 Nov 3;375(18):1738-1748. doi: 10.1056/NEJMoa1609709. Epub 2016 Oct 7. PMID 27717303
- [Background] Hortobagyi GN, Stemmer SM, Burris HA, Yap YS, Sonke GS, Paluch-Shimon S, Campone M, Petrakova K, Blackwell KL, Winer EP, Janni W, Verma S, Conte P, Arteaga CL, Cameron DA, Mondal S, Su F, Miller M, Elmeliegy M, Germa C, O'Shaughnessy J. Updated results from MONALEESA-2, a phase III trial of first-line ribociclib plus letrozole versus placebo plus letrozole in hormone receptor-positive, HER2-negative advanced breast cancer. Ann Oncol. 2018 Jul 1;29(7):1541-1547. doi: 10.1093/annonc/mdy155. PMID 29718092
- [Background] Swain SM, Miles D, Kim SB, Im YH, Im SA, Semiglazov V, Ciruelos E, Schneeweiss A, Loi S, Monturus E, Clark E, Knott A, Restuccia E, Benyunes MC, Cortes J; CLEOPATRA study group. Pertuzumab, trastuzumab, and docetaxel for HER2-positive metastatic breast cancer (CLEOPATRA): end-of-study results from a double-blind, randomised, placebo-controlled, phase 3 study. Lancet Oncol. 2020 Apr;21(4):519-530. doi: 10.1016/S1470-2045(19)30863-0. Epub 2020 Mar 12. PMID 32171426
- [Background] Andre F, Ciruelos E, Rubovszky G, Campone M, Loibl S, Rugo HS, Iwata H, Conte P, Mayer IA, Kaufman B, Yamashita T, Lu YS, Inoue K, Takahashi M, Papai Z, Longin AS, Mills D, Wilke C, Hirawat S, Juric D; SOLAR-1 Study Group. Alpelisib for PIK3CA-Mutated, Hormone Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2019 May 16;380(20):1929-1940. doi: 10.1056/NEJMoa1813904. PMID 31091374
- [Background] Di Leo A, Jerusalem G, Petruzelka L, Torres R, Bondarenko IN, Khasanov R, Verhoeven D, Pedrini JL, Smirnova I, Lichinitser MR, Pendergrass K, Garnett S, Lindemann JP, Sapunar F, Martin M. Results of the CONFIRM phase III trial comparing fulvestrant 250 mg with fulvestrant 500 mg in postmenopausal women with estrogen receptor-positive advanced breast cancer. J Clin Oncol. 2010 Oct 20;28(30):4594-600. doi: 10.1200/JCO.2010.28.8415. Epub 2010 Sep 20. PMID 20855825
- [Background] Di Leo A, Johnston S, Lee KS, Ciruelos E, Lonning PE, Janni W, O'Regan R, Mouret-Reynier MA, Kalev D, Egle D, Csoszi T, Bordonaro R, Decker T, Tjan-Heijnen VCG, Blau S, Schirone A, Weber D, El-Hashimy M, Dharan B, Sellami D, Bachelot T. Buparlisib plus fulvestrant in postmenopausal women with hormone-receptor-positive, HER2-negative, advanced breast cancer progressing on or after mTOR inhibition (BELLE-3): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2018 Jan;19(1):87-100. doi: 10.1016/S1470-2045(17)30688-5. Epub 2017 Dec 7. PMID 29223745
- [Background] Sammons S, Kornblum NS, Blackwell KL. Fulvestrant-Based Combination Therapy for Second-Line Treatment of Hormone Receptor-Positive Advanced Breast Cancer. Target Oncol. 2019 Feb;14(1):1-12. doi: 10.1007/s11523-018-0587-9. PMID 30136059
- [Background] Murthy RK, Loi S, Okines A, Paplomata E, Hamilton E, Hurvitz SA, Lin NU, Borges V, Abramson V, Anders C, Bedard PL, Oliveira M, Jakobsen E, Bachelot T, Shachar SS, Muller V, Braga S, Duhoux FP, Greil R, Cameron D, Carey LA, Curigliano G, Gelmon K, Hortobagyi G, Krop I, Loibl S, Pegram M, Slamon D, Palanca-Wessels MC, Walker L, Feng W, Winer EP. Tucatinib, Trastuzumab, and Capecitabine for HER2-Positive Metastatic Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):597-609. doi: 10.1056/NEJMoa1914609. Epub 2019 Dec 11. PMID 31825569
- [Background] Bredin P, Walshe JM, Denduluri N. Systemic therapy for metastatic HER2-positive breast cancer. Semin Oncol. 2020 Oct;47(5):259-269. doi: 10.1053/j.seminoncol.2020.07.008. Epub 2020 Aug 18. PMID 32896428
- [Background] Zhao W, Bian L, Wang T, Zhang S, Li J, Xu F, Jiang Z. Effectiveness of second-line anti-HER2 treatment in HER2-positive metastatic breast cancer patients previously treated with trastuzumab: A real-world study. Chin J Cancer Res. 2020 Jun;32(3):361-369. doi: 10.21147/j.issn.1000-9604.2020.03.07. PMID 32694900
- [Background] Kelly P, Ma Z, Baidas S, Moroose R, Shah N, Dagan R, Mamounas E, Rineer J. Patterns of Progression in Metastatic Estrogen Receptor Positive Breast Cancer: An Argument for Local Therapy. Int J Breast Cancer. 2017;2017:1367159. doi: 10.1155/2017/1367159. Epub 2017 Sep 25. PMID 29147583
- [Background] Weickhardt AJ, Scheier B, Burke JM, Gan G, Lu X, Bunn PA Jr, Aisner DL, Gaspar LE, Kavanagh BD, Doebele RC, Camidge DR. Local ablative therapy of oligoprogressive disease prolongs disease control by tyrosine kinase inhibitors in oncogene-addicted non-small-cell lung cancer. J Thorac Oncol. 2012 Dec;7(12):1807-1814. doi: 10.1097/JTO.0b013e3182745948. PMID 23154552
- [Background] Cheung P, Patel S, North SA, Sahgal A, Chu W, Soliman H, Ahmad B, Winquist E, Niazi T, Patenaude F, Lim G, Heng DYC, Dubey A, Czaykowski P, Wong RKS, Swaminath A, Morgan SC, Mangat R, Keshavarzi S, Bjarnason GA. Stereotactic Radiotherapy for Oligoprogression in Metastatic Renal Cell Cancer Patients Receiving Tyrosine Kinase Inhibitor Therapy: A Phase 2 Prospective Multicenter Study. Eur Urol. 2021 Dec;80(6):693-700. doi: 10.1016/j.eururo.2021.07.026. Epub 2021 Aug 13. PMID 34399998
- [Background] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Background] Hannan R, Christensen M, Hammers H, Christie A, Paulman B, Lin D, Garant A, Arafat W, Courtney K, Bowman I, Cole S, Sher D, Ahn C, Choy H, Timmerman R, Brugarolas J. Phase II Trial of Stereotactic Ablative Radiation for Oligoprogressive Metastatic Kidney Cancer. Eur Urol Oncol. 2022 Apr;5(2):216-224. doi: 10.1016/j.euo.2021.12.001. Epub 2022 Jan 2. PMID 34986993
- [Background] Yu HA, Sima CS, Huang J, Solomon SB, Rimner A, Paik P, Pietanza MC, Azzoli CG, Rizvi NA, Krug LM, Miller VA, Kris MG, Riely GJ. Local therapy with continued EGFR tyrosine kinase inhibitor therapy as a treatment strategy in EGFR-mutant advanced lung cancers that have developed acquired resistance to EGFR tyrosine kinase inhibitors. J Thorac Oncol. 2013 Mar;8(3):346-51. doi: 10.1097/JTO.0b013e31827e1f83. PMID 23407558
- [Background] Tsai CJ, Yang JT, Guttmann DM et al. Consolidative Use of Radiotherapy to Block (CURB) Oligoprogression - Interim Analysis of the First Randomized Study of Stereotactic Body Radiotherapy in Patients With Oligoprogressive Metastatic Cancers of the Lung and Breast, Int J Radiat Oncol Biol Phys. 2021; 111(5):1325-1326.
- [Background] Triggiani L, Alongi F, Buglione M, Detti B, Santoni R, Bruni A, Maranzano E, Lohr F, D'Angelillo R, Magli A, Bonetta A, Mazzola R, Pasinetti N, Francolini G, Ingrosso G, Trippa F, Fersino S, Borghetti P, Ghirardelli P, Magrini SM. Efficacy of stereotactic body radiotherapy in oligorecurrent and in oligoprogressive prostate cancer: new evidence from a multicentric study. Br J Cancer. 2017 Jun 6;116(12):1520-1525. doi: 10.1038/bjc.2017.103. Epub 2017 Apr 27. PMID 28449007
- [Background] Alomran R, White M, Bruce M, Bressel M, Roache S, Karroum L, Hanna GG, Siva S, Goel S, David S. Stereotactic radiotherapy for oligoprogressive ER-positive breast cancer (AVATAR). BMC Cancer. 2021 Mar 23;21(1):303. doi: 10.1186/s12885-021-08042-w. PMID 33757458
- [Background] Tan H, Cheung P, Louie AV, Myrehaug S, Niglas M, Atenafu EG, Chu W, Chung HT, Poon I, Sahgal A, Soliman H. Outcomes of extra-cranial stereotactic body radiotherapy for metastatic breast cancer: Treatment indication matters. Radiother Oncol. 2021 Aug;161:159-165. doi: 10.1016/j.radonc.2021.06.012. Epub 2021 Jun 10. PMID 34119585
- [Background] Weykamp F, Konig L, Seidensaal K, Forster T, Hoegen P, Akbaba S, Mende S, Welte SE, Deutsch TM, Schneeweiss A, Debus J, Horner-Rieber J. Extracranial Stereotactic Body Radiotherapy in Oligometastatic or Oligoprogressive Breast Cancer. Front Oncol. 2020 Jun 26;10:987. doi: 10.3389/fonc.2020.00987. eCollection 2020. PMID 32676455
- [Background] Donovan E, Dhesy-Thind S, Mukherjee S, Kucharczyk M, Swaminath A. Attitudes and beliefs toward the use of stereotactic body radiotherapy in oligometastatic breast cancer: A commentary on a survey of Canadian Medical Oncologists. Breast J. 2019 Nov;25(6):1222-1224. doi: 10.1111/tbj.13435. Epub 2019 Jul 1. PMID 31264272
- [Background] Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. US Department of Health, National Institutes of Health and National Cancer Institude. 2017. Published online: https://academy.myeloma.org.uk/wp-content/uploads/2015/04/CTCAE_v5.pdf
- [Background] Timmerman R. A Story of Hypofractionation and the Table on the Wall. Int J Radiat Oncol Biol Phys. 2022 Jan 1;112(1):4-21. doi: 10.1016/j.ijrobp.2021.09.027. No abstract available. PMID 34919882
- [Background] Sahgal A, Myrehaug SD, Siva S, Masucci L, Foote MC, Brundage M, Butler J, Chow E, Fehlings MG, Gabos Z, Greenspoon J, Kerba M, Lee YK, Liu MC, Maralani P, Thibault I, Wong R, Hum M, Ding K, Parulekar W. CCTG SC.24/TROG 17.06: A Randomized Phase II/III Study Comparing 24Gy in 2 Stereotactic Body Radiotherapy (SBRT) Fractions Versus 20Gy in 5 Conventional Palliative Radiotherapy (CRT) Fractions for Patients with Painful Spinal Metastases. Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1397-1398. doi: 10.1016/j.ijrobp.2020.09.019. Epub 2020 Nov 18. No abstract available. PMID 33427654
- [Background] Response assessment in solid tumors (RECIST):Version 1.1 and Supporting Papers. European Journal of Cancer. 2009. 45 (2): 225-310.